CLINICAL TRIAL: NCT05657301
Title: A Phase I, Open-label, Multicenter, Dose-Escalating Study to Evaluate the Safety and Tolerability of KH631 Gene Therapy in Participants With Neovascular Age-related Macular Degeneration
Brief Title: Safety and Tolerability of KH631 Gene Therapy in Participants With Neovascular Age-related Macular Degeneration
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Origen Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chengdu Kanghong Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAN-2201
Record Dates: First submitted 2022-12-10; First posted 2022-12-20 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- KH631 Dose 1 (Experimental): KH631 One-Time Intraocular Injection Dose Level 1
  Interventions: Drug: KH631
- KH631 Dose 2 (Experimental): KH631 One-Time Intraocular Injection Dose Level 2
  Interventions: Drug: KH631
- KH631 Dose 3 (Experimental): KH631 One-Time Intraocular Injection Dose Level 3
  Interventions: Drug: KH631
- KH631 Dose 4 (Experimental): KH631 One-Time Intraocular Injection Dose Level 4
  Interventions: Drug: KH631
- KH631 Dose 5 (Experimental): KH631 One-Time Intraocular Injection Dose Level 5
  Interventions: Drug: KH631

INTERVENTIONS:
Drug: KH631 — KH631: AAV vector containing a coding sequence for an anti-VEGF protein

SUMMARY:
VAN-2201 is Phase I clinical trial to assess the safety and tolerability of KH631 in subjects with neovascular AMD. KH631 is gene therapy designed to deliver a protein which targets and blocks VEGF via an adeno-associated viral vector. The standard of care for patients with neovascular AMD are anti-VEGF treaments, which have demonstrated improvement in vision and reduction in fluid. A one time placement of a product which inhibits VEGF has the potential to reduce the patient burden of regular intraocular injections.

DETAILED DESCRIPTION:
The VAN-2201 clinical trial is a multicenter, open-label, dose-escalating clinical study. The primary objective of the study will be to establish a safe and tolerable dose range in subjects with neovascular AMD. Five dose cohorts are planned to be included in the study, with approximately five subjects per cohort. Subjects who meet the eligibility criteria (i.e. all the inclusion and no exclusion criteria) will be enrolled to receive KH631. KH631 will be delivered at the dose level according to the cohort via intraocular injection. Subjects will be seen monthly until the primary outcome measurement at 24 weeks and through week 52. The subjects will be continued to followed with regular visits until they complete the 104 week visit.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females ages 50 to 85 (inclusive) with a study eye which meets the following criteria:

a. Previously received IVT treatment of anti-VEGF for neovascular AMD, with documented response to anti-VEGF therapy during the first 2 weeks of screening b. active macular CNV lesion secondary to AMD evidenced by SD-OCT c. Have a ETDRS BCVA letter score of 63 to 19 (approximately 20/63 to 20/400 Snellen equivalent) in the study eye at Screening for the first subject in each cohort (sentinel subject), followed by ETDRS BCVA letter score of 73 to 19 (approximately 20/40 to 20/400 Snellen equivalent) for the rest of the subjects each cohort; d. Pseudophakia in the study eye, with ocular media to permit high quality fundus imaging at screening and allow planned vitrectomy and subretinal injection; e. Are willing and able to sign the study written informed consent form (ICF).

Exclusion Criteria:

1. Have had any prior ocular or systemic treatment (investigational or approved) or surgery for the treatment of neovascular AMD except IVT anti-VEGF
2. Retinal pigment epithelial tears or rips at screening
3. Any history or presence of vitreous hemorrhage;
4. Have any condition preventing visual acuity improvement;
5. Have any other cause of CNV; prior pars plana vitrectomy or scleral buckling or retinal detachment surgery; macular hole, Epiretinal membrane or vitreo-macular traction; full thickness macular hole;
6. History of intraocular or periocular surgery in the prior 3 months;
7. Prior trabeculectomy or other filtration surgery ;
8. Any use of long-acting intraocular steroids, including implants, within six months prior;

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Safety (Type, Severity and Incidence of ocular and systemic AEs and SAEs) | 52 Weeks
  type, severity and incidence of ocular and systemic AEs and SAEs
Best Corrected Visual Acuity | 52 Weeks
  Change in Best Corrected Visual Acuity

SECONDARY OUTCOMES:
Safety (type, severity and incidence of ocular and systemic AEs and SAEs) | 104 Weeks
  type, severity and incidence of ocular and systemic AEs and SAEs
Rescue Injections | 104 Weeks
  Mean Number of Rescue Injections
Best Corrected Visual Acuity | 104 Weeks
  Change in Best Corrected Visual Acuity

CONTACTS AND LOCATIONS:
Overall Officials: Avner Ingerman, MD, MSc, Study Director — Vanotech Ltd.
Locations (7):
- United States (7):
  - Kanghong Investigative Site, Phoenix, Arizona
  - Kanghong Investigative Site, Lemont, Illinois
  - Kanghong Investigative Site, Boston, Massachusetts
  - Kanghong Investigative Site, Reno, Nevada
  - Kanghong Investigative Site, Cherry Hill, New Jersey
  - Kanghong Investigative Site, Germantown, Tennessee
  - Kanghong Investigative Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No